CLINICAL TRIAL: NCT05539846
Title: Optimization and Effect Analysis of Blood Collection Method Based on Patient Demand
Brief Title: Explore the Feasibility of Modified Blood Collection Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xin Fu, Director, Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TZhospital 001
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Autologous Blood Transfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental)
  Interventions: Procedure: modified blood collection method
- control group (No Intervention)

INTERVENTIONS:
Procedure: modified blood collection method — The bevel of the needle head of the blood collection needle was downward, and the needle was inserted into the skin with the bevel of the needle parallel to the skin.
  Arms: test group

SUMMARY:
Blood collection method: routine preparation according to predeposit autologous blood transfusion. Control group: according to the conventional blood collection method, the bevel of the needle head of the blood collection needle was upward, and the needle was inserted at an angle of 30-45 degrees according to the patient's blood vessel. Test group: the bevel of the needle head of the blood collection needle was downward, and the needle was inserted into the skin with the bevel of the needle parallel to the skin. The other blood collection operations of the two groups were the same, the blood collection volume was 400 mL and the routine treatment was performed after the blood collection. Blood collection process was as follows.

1. Check the patient information and prepare for blood collection.
2. Explain the purpose, significance and operation process to the patients, get the understanding of the patients and their families, and sign the informed consent.
3. Close the doors and windows, pull the bed curtain, pay attention to protect the patient's privacy, and the patient should wear a mask.
4. Assist the patient to take the flat lying position, select the middle elbow vein, and strictly disinfect the local skin. In the control group, the wedge-shaped slope of the needle head of the blood collection needle is upward, and the needle is inserted at an angle of 30-45 degrees according to the blood vessel condition of the patient. In the experimental group, the wedge-shaped slope of the needle head of the blood collection needle is downward, and the needle is inserted parallel to the skin. After the puncture is successful, shake the blood bag evenly to prevent hemolysis and blood clot.
5. The nurse shall first establish a venous access (standby) for the patient on the opposite limb of the blood collection, measure the patient's blood pressure and pulse and record it, and give ECG monitoring if necessary. During blood collection, observe the patient's complexion and pulse, and ask if there are symptoms such as palpitation, chest tightness and chest pain. The patient with ECG monitoring shall pay attention to the heart rhythm and heart rate.
6. When the blood collection reaches the predetermined blood volume, pull out the needle and compress the needle eye with a dry cotton ball for 5 ~ 10 minutes. Especially in older patients, bleeding should be prevented due to poor vascular elasticity. The blood bag drainage tube shall be sealed with a hot press sealing machine, and the patient's name, hospitalization number, blood type, blood volume, blood collection date, blood collector and nurse's signature shall be indicated. It shall be sent to the blood bank for storage at 4 ℃, and the effective storage period is 21 days. The patient's blood pressure and pulse were measured again and recorded.
7. The blood was collected 1 ~ 2 weeks before operation, and can be stored for 1 ~ 3 times. Each time the blood collection volume was 10 ml / kg body weight. The interval between the two blood storage was about 3 days. The blood storage was stopped 3 days before operation.
8. Record all indicators. The size of bruises (spots) was measured after 24 hours.

Observation indicators: ① blood spilled from the bevel of the needle when the needle was inserted; ② the diameter of the bruise area was greater than 5 mm after 24 hours; ③ there was a blood clot during the autologous blood transfusion when checked; ④ changes of heart rate and blood pressure before and after blood collection; ⑤ patient pain score (NRS score); ⑥ time required to collect 400 ml of blood; ⑦ adverse reactions, dizziness, palpitations, pale complexion, low volume shock, etc.

Statistical methods: SPSS 25.0 statistical software was used for statistical analysis of the data. The measurement data were subject to normal distribution and expressed by mean ± standard deviation (). Independent sample t-test was used for inter group comparison. Paired sample t-test was used for comparison before and after treatment. The counting data was expressed by rate or constituent ratio (%), and chi square test was used for inter group comparison (χ2), inspection level α=0.05。

ELIGIBILITY:
Inclusion Criteria:

* weight: ≥50 Kg;
* hemoglobin ≥110 g/L;
* heart function: I-II;
* patients who were expected to have a large amount of surgical bleeding and might require blood transfusion;
* with surgical indications and surgical conditions.

Exclusion Criteria:

* having a history of hematophobia;
* having communication difficulties and cannot cooperate;
* having blood collection interruption caused by various accidents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
incidence of blood spill | when the needle was inserted
  The incidence of blood spill of the control group is 80.9%, while it of the test group is 0.00%.
incidence of bruise area | after 24 hours
  The incidence of bruise area of the control group is 63.8%, while it of the test group is 13.3%.
incidence of blood clot | during the autologous blood transfusion when checked
  The incidence of blood clot of the control group is 10.6%, while it of the test group is 0.00%.
incidence of dizziness | After blood collection
  The incidence of dizziness of the control group is 2.1%, while it of the test group is 2.2%.
heart rate | before and after blood collection
  Heart rate of the control group before and after blood collection is 77.19±6.20 and 77.94±6.83 respectively. Heart rate of the test group before and after blood collection is 76.11±5.59 and 77.22±4.32 respectively.
blood pressure | before and after blood collection
  Systolic blood pressure of the control group before and after blood collection is 124.85±7.94 and 125.7±6.75 respectively. Systolic blood pressure of the test group before and after blood collection is 124.93±7.04 and 125.76±6.41 respectively. Diastolic blood pressure of the control group before and after blood collection is 77.87±5.79 and 77.43±4.29 respectively. Diastolic blood pressure of the test group before and after blood collection is 77.62±5.08 and 76.6±4.40 respectively.
patient pain score | during blood collection
  Patient pain score of the control group is 12.51±0.98. Patient pain score of the test group is 1.53±0.69.
the time required to collect 400 mL of blood | during blood collection
  The time required to collect 400 mL of blood of the control group is 766.62±83.18. The time required to collect 400 mL of blood of the test group is 481.98±69.76.

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia L, Wang Y, Zhang W, Lin Y, Chen F, Wan Y, Fu X. Optimisation and Effect Analysis of the Blood Collection Method in Pre-Deposit Autotransfusion Patients Undergoing Thoracotomy Surgery. J Multidiscip Healthc. 2023 Sep 20;16:2793-2798. doi: 10.2147/JMDH.S424470. eCollection 2023. PMID 37753340